CLINICAL TRIAL: NCT07400302
Title: A Randomized, Controlled, Multicenter Phase II Clinical Study Evaluating the Adjuvant Treatment of PD-L1-Positive, Resectable Mucosal Melanoma With Sintilimab Plus Chemotherapy Versus Chemotherapy Alone
Brief Title: Sintilimab Combined With Chemotherapy for Adjuvant Treatment of Mucosal Melanoma After Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K2024390
Record Dates: First submitted 2026-01-21; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-02

CONDITIONS: Mucosal Melanoma; PD-L1 Positive
Keywords: Adjuvant Treatment; PD-L1-Positive; Resectable Mucosal Melanoma; immunotherapy
MeSH Terms: interventions — sintilimab; Dacarbazine; Temozolomide; Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group A (Experimental): Sintilimab, Dacarbazine or Temozolomide, Combined with Cisplatin
  Interventions: Drug: Sintilimab; Drug: Dacarbazine or Temozolomide; Drug: Cisplatin
- Experimental group B (Active Comparator): Dacarbazine or Temozolomide, Combined with Cisplatin
  Interventions: Drug: Dacarbazine or Temozolomide; Drug: Cisplatin

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200 mg IV Q3W for 6 cycles. Followed by maintenance therapy with sintilimab 200 mg IV Q3W for 1 year.
  Arms: Experimental group A
Drug: Dacarbazine or Temozolomide — Dacarbazine 250 mg/m² or Temozolomide 200 mg/m² QD D1-5 Q3W for 6 cycles.
Drug: Cisplatin — Cisplatin 75 mg/m² IV D1-3 Q3W, administered in combination for 6 cycles.

SUMMARY:
Melanoma has emerged as the fastest-growing malignancy in recent years, with incidence and mortality rates among both men and women in East Asian countries exceeding the Asian average. China ranks fifth among East Asian nations in melanoma incidence. Currently, immune checkpoint inhibitors are achieving significant breakthroughs in adjuvant melanoma therapy. This study aims to evaluate the efficacy and safety of sintilimab combined with chemotherapy versus chemotherapy alone in patients with PD-L1-positive, completely resectable mucosal melanoma, thereby providing additional clinical evidence for treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form (Informed Consent, ICF) and be able to comply with the visit schedule and related procedures outlined in the protocol.
2. Histologically/cytologically confirmed mucosal melanoma, with primary and/or metastatic lesions completely resected, with negative surgical margins.
3. Tissue specimen: PD-L1 positive (CPS ≥ 1).
4. The first dose of the study drug must be administered only after the melanoma resection wound has fully healed, and the injection time must not exceed 13 weeks post-surgery (if the time limit is exceeded by no more than 7 days due to unforeseen circumstances, the decision to enroll may be discussed with the medical monitor).
5. Confirmed R0 complete resection by physical examination and imaging within 4 weeks prior to randomization.
6. For central nervous system (CNS) metastasis, post-surgical resection may receive adjuvant radiotherapy as needed. MRI of the brain must show no recurrence for at least 4 weeks after surgery or surgery combined with radiotherapy. Note: if immunosuppressants (e.g., prednisone) are required, they must be discontinued at least 14 days before the study drug administration.
7. If lymph node dissection combined with local radiotherapy is required after melanoma resection, radiotherapy must be completed within 13 weeks of lymph node dissection and before the start of adjuvant treatment. Note: If delayed wound healing occurs due to radiotherapy, the subject will not meet the eligibility criteria.
8. Age ≥ 18 years.
9. Expected survival ≥ 12 weeks.
10. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
11. Sufficient organ and bone marrow function, with laboratory values meeting the following criteria within 7 days before enrollment (no blood components, cell growth factors, albumin, or other intravenous or subcutaneous corrective drugs should be given within 14 days prior to laboratory tests):

(1) Hematology: Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L; Platelet Count (PLT) ≥ 90 × 10⁹/L; Hemoglobin (HGB) ≥ 9.0 g/dL (90 g/L).

(2) Liver Function: Total Bilirubin (TBIL) ≤ 1.5 × the upper limit of normal (ULN) (for patients suspected of or diagnosed with Gilbert's syndrome, TBIL ≤ 3 × ULN); Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 × ULN.

(3) Renal Function: Serum Creatinine (Scr) ≤ 1.5 × ULN, or Creatinine Clearance Rate (Ccr) ≥ 50 ml/min (calculated using the Cockcroft/Gault formula), and urinalysis showing urinary protein (UPRO) < 2+ or 24-hour urinary protein < 1g.(Cockcroft-Gault Formula) (4) Coagulation Function: International Normalized Ratio (INR) and Prothrombin Time (PT) ≤ 1.5 × ULN.

12. Female subjects of childbearing potential, or male subjects whose partners are women of childbearing potential, must use effective contraception throughout the treatment period and for 6 months after treatment.

Exclusion Criteria:

1. Previous exposure to any anti-PD-1 or anti-PD-L1/2 antibody.
2. Previous use of interferon.
3. Hyperthyroidism or hypothyroidism. Note: Hypothyroid patients whose condition is stable after hormone replacement therapy may be included.
4. Concurrent participation in another clinical trial.
5. Receipt of any investigational drug within 4 weeks before the first dose of the study drug.
6. Use of immunosuppressive drugs within 4 weeks prior to the first dose of the study drug, excluding nasal, inhaled, or other topical corticosteroids or systemic corticosteroids at physiological doses (i.e., not exceeding 10 mg/day of prednisone or an equivalent dose of other corticosteroids).
7. Receipt of live attenuated vaccines within 4 weeks before the first dose of the study drug or planned use during the study.
8. Major surgery (e.g., craniotomy, thoracotomy, or laparotomy) or any unhealed wounds, ulcers, or fractures within 4 weeks before the first dose of the study drug.
9. History of gastrointestinal perforation and/or fistulas within 6 months prior to the first dose of the study drug.
10. Previous systemic anticancer treatment (e.g., chemotherapy, targeted therapy, or biologics). Chinese herbal medicine with anticancer indications or immunomodulatory drugs (e.g., thymosin, interleukins) are allowed after a 2-week washout period.
11. Active, known, or suspected autoimmune diseases, or a history of autoimmune disease within the last 2 years (subjects with vitiligo, psoriasis, alopecia, or Grave's disease who did not require systemic treatment in the past 2 years, hypothyroidism requiring only thyroid hormone replacement therapy, and type 1 diabetes requiring only insulin replacement therapy may be included).
12. Known history of primary immunodeficiency.
13. Known history of organ transplantation (except corneal transplant) or hematopoietic stem cell transplant.
14. History of idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-induced pneumonia, or any pulmonary diseases with severe impairment of lung function.
15. Known history of severe allergic reactions to other monoclonal antibodies or interferons, or to any ingredient in the study drug (e.g., sintilimab or interferon).
16. Clinically uncontrolled third-space fluid accumulation, such as pleural effusion or ascites that cannot be controlled by drainage or other methods before enrollment.
17. HIV infection (HIV antibody positive).
18. Acute or chronic active hepatitis B (HBV DNA copy number ≥ 1 × 10³ copies/ml or ≥ 200 IU/ml) or acute or chronic active hepatitis C (HCV antibody positive); patients with HCV antibody positive but RNA negative are eligible for inclusion.
19. Active pulmonary tuberculosis.
20. Active or clinically uncontrolled severe infections.
21. Symptomatic congestive heart failure (NYHA Class III-IV) or symptomatic or uncontrolled arrhythmia.
22. Uncontrolled hypertension despite appropriate treatment (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).
23. Any arterial thromboembolic event (e.g., myocardial infarction, unstable angina, pulmonary embolism, cerebral embolism) within 6 months before enrollment.
24. History of deep vein thrombosis or any other severe thromboembolic event within 3 months before enrollment (implanted venous infusion ports or catheter-related thrombosis or superficial vein thrombosis are not considered "severe" thromboembolic events).
25. Uncontrolled metabolic disorders or other non-malignant organ/systemic diseases or cancer sequelae that would increase medical risks and/or create uncertainties in survival prognosis, and the investigator judges that the patient is unsuitable for enrollment.
26. Hepatic encephalopathy, hepatorenal syndrome, or decompensated cirrhosis (Child-Pugh Class B or C).
27. History of gastrointestinal perforation and/or fistulae, bowel obstruction (including incomplete bowel obstruction requiring parenteral nutrition), extensive bowel resection (e.g., partial colon or extensive small bowel resection resulting in chronic diarrhea), Crohn's disease, ulcerative colitis, or long-term chronic diarrhea within 6 months prior to enrollment.
28. Other acute or chronic diseases, psychiatric disorders, or abnormal laboratory test results that may:

(1) Increase the risk related to participation in the study or study drug administration.

(2) Interfere with the interpretation of study results and lead the investigator to determine that the patient is ineligible for participation.

29. History of other primary malignancies, excluding:

1. Malignancies that have been cured with no evidence of active disease for at least 5 years prior to enrollment, with a very low risk of recurrence.
2. Non-melanoma skin cancer or malignant lentigo maligna with no evidence of disease recurrence after sufficient treatment.
3. In situ carcinoma that has been treated sufficiently with no evidence of recurrence.

30. Pregnant or breastfeeding female patients. 31. Other conditions that, according to the investigator's judgment, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | 2 years

SECONDARY OUTCOMES:
2-year recurrence-free survival rate | 2 years
Overall Survival | 3 years
  Time from randomization to documented death from any cause.
Number of participants with treatment-emergent adverse events (TEAEs) as assessed by CTCAE v5.0. | From the first dose of study treatment up to 30 days after the last dose.
  Safety will be assessed in the Safety Set (SS), including all participants who received at least one dose of study medication. Assessments include the incidence and severity of adverse events, laboratory abnormalities (hematology, liver/kidney function), vital signs, ECG changes, and immunogenicity.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No